CLINICAL TRIAL: NCT06243679
Title: The Efficacy and Safety of Adjuvant Immunotherapy After Pathological Complete Response Following Neoadjuvant Chemoimmunotherapy in Patients with Resectable NSCLC: a Prospective Real-World Study
Brief Title: The Efficacy and Safety of Adjuvant Immunotherapy After Pathological Complete Response Following Neoadjuvant Chemoimmunotherapy in Patients with Resectable NSCLC
Status: Active, not recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: RWNEOADJ-01
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-01

CONDITIONS: Resectable/Potentially Resectable NSCLC
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adjuvant immunotherapy
  Interventions: Drug: Immunotherapy
- Observational

INTERVENTIONS:
Drug: Immunotherapy — Monotherapy with PD-1 inhibitors, up to 1 year.
  Groups: Adjuvant immunotherapy

SUMMARY:
This is a prospective, observational, multicenter real-world study aiming to investigate the efficacy and safety of NSCLC patients with or without adjuvant immunotherapy who have achieved pathologic complete remission after neoadjuvant immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years ≤ age ≤ 80 years;
2. Histologically or cytologically confirmed NSCLC;
3. Resectable stage IB, II, IIIA, or IIIB (N2) NSCLC according to the staging criteria of the American Joint Committee on Cancer (8th edition);
4. Eastern Cooperative Oncology Group (ECOG) performance status score 0-1 at baseline;
5. With measurable or evaluable diseases according to the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) at baseline;
6. Achieving pathological complete response (pCR) after three cycles of neoadjuvant chemoimmunotherapy, which was assessed by independent pathological examination of surgical specimens;
7. With or without adjuvant immunotherapy postoperatively;
8. Signed and dated written informed consent provided by the patient prior to admission to the study.

Exclusion Criteria:

1. EGFR or ALK aberrations positive;
2. With primary/secondary immunodeficiency diseases or symptomatic interstitial lung diseases;
3. With a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days of study drug administration;
4. With other active malignant tumors currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drugs;
5. Receipt of other investigational drugs during the observation period;
6. Unable to follow the procedures required in the protocol due to any medical, mental or psychological conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with resectable non-small cell lung cancer (NSCLC) who have received immune checkpoint inhibitor neoadjuvant therapy and achieved pathological complete response (pCR).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
DFS (Disease-Free Survival) | Approximately 3 years
  Evaluated by investigator based on RECIST1.1

SECONDARY OUTCOMES:
3-year DFS (disease-free survival) rate | Approximately 3 years
  Evaluated by investigator based on RECIST1.1
OS (Overall Survival) | Approximately 3 years
  Evaluated by investigator based on RECIST1.1
Recurrence and Metastasis Pattern | Approximately 3 years
AE (Adverse Event) | Approximately 3 years
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered an investigational product. Safety and tolerance evaluated by incidence, severity and outcomes of AEs (according to NCICTCAE 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University Affiliated, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No